CLINICAL TRIAL: NCT04621526
Title: Monitored Anesthesia Care: Dexmedetomidine-Ketamine Versus Dexmedetomidine- Propofol Combination During Burr-Hole Surgery For Chronic Subdural Hematoma
Brief Title: Monitored Anesthesia Care: Dexmedetomidine-Ketamine Versus Dexmedetomidine- Propofol For Chronic Subdural Hematoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Alshaimaa Abdel Fattah Kamel, principle investigator, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 6434
Record Dates: First submitted 2020-10-28; First posted 2020-11-09 (Actual); Last update posted 2023-10-17 (Actual); Status verified 2023-10

CONDITIONS: Conscious Sedation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- dexmedetomidine- ketamine (Active Comparator): patients will receive combination of ketamine 1mg/kg and dexmedetomidine 1ug/kg diluted in 10 ml 0.9% saline infused over 10 min together as an intravenous bolus dose then a maintenance of 0.5ug/kg/h dexmedetomidine and ketamine 0.5 mg/kg/h continuous infusion in two separate syringes pump to achieve modified Observer's Assessment of Alertness and sedation score (OAA/S) 3 and the infusion will stopped by finishing the skin suture.
  Interventions: Drug: dexmedetomidine- ketamine
- dexmedetomidine- propofol (Active Comparator): patients will receive combination from 1 mg/kg propofol and dexmedetomidine 1ug/kg diluted in 10 ml 0.9% saline infused over 10 min together as an intravenous bolus dose then a maintenance of 0.5ug/kg/h dexmedetomidine and propofol 1 mg/kg/h continuous infusion in two separate syringes pump to achieve modified Observer's Assessment of Alertness and sedation score (OAA/S) 3 and the infusion will stopped by finishing the skin suture.
  Interventions: Drug: dexmedetomidine- propofol

INTERVENTIONS:
Drug: dexmedetomidine- ketamine — patients will receive combination of ketamine 1mg/kg and dexmedetomidine 1ug/kg diluted in 10 ml 0.9% saline infused over 10 min together as an intravenous bolus dose then a maintenance of 0.5ug/kg/h dexmedetomidine and ketamine 0.5 mg/kg/h continuous infusion in two separate syringes pump to achieve modified Observer's Assessment of Alertness and sedation score (OAA/S) 3 and the infusion will stopped by finishing the skin suture.
  Other Names: precedex- katalar
  Arms: dexmedetomidine- ketamine
Drug: dexmedetomidine- propofol — patients will receive combination from 0.5 mg/kg propofol and dexmedetomidine 1ug/kg diluted in 10 ml 0.9% saline infused over 10 min together as an intravenous bolus dose then a maintenance of 0.5ug/kg/h dexmedetomidine and propofol 0.5 mg/kg/h continuous infusion in two separate syringes pump to achieve modified Observer's Assessment of Alertness and sedation score (OAA/S) 3 and the infusion will stopped by finishing the skin suture.
  Other Names: precedex- diprivan
  Arms: dexmedetomidine- propofol

SUMMARY:
Inadequate sedation and analgesia indicated by intraoperative movements are markers of inadequate MAC during burr-hole surgery for chronic subdural hematoma evacuation especially when general anesthesia poses high risk for the patients.

Dexmedetomidine, ketamine, propofol intravenous infusion and other agents was used to provide monitored anesthesia care with variable success if used as solitary agents as each drug has its limited use.

DETAILED DESCRIPTION:
* Null hypothesis (H0): There are no differences between the effects of dexmedetomidine- ketamine and dexmedetomidine- propofol combination for monitored anesthesia care during burr-hole surgery for chronic subdural hematoma evacuation.
* Alternative hypothesis (H1): There are differences between the effects of dexmedetomidine- ketamine and dexmedetomidine- propofol combination for monitored anesthesia care during burr-hole surgery for chronic subdural hematoma evacuation.

ELIGIBILITY:
Inclusion Criteria:

* Patient acceptance.
* Both sex.
* Age (50-80) years old.
* Patient with Body Mass Index (BMI) (25-30kg/m²).
* American Society of Anesthesiologist (ASA) II / III
* patient scheduled to burr-hole surgery for chronic subdural hematoma evacuation under MAC.

Exclusion Criteria:

* Patient with difficult airway (mallapati III,IV).
* Altered mental status (psychiatric and anexity disorder).
* Post-traumatic stress disorders.
* History of allergy to study drugs.
* Patient on sedative or hypnotic medication.
* Patients with on painkiller.
* Patients with any degree of heart block.
* Sever liver, respiratory or renal impairment.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2020-11-10 (Actual); Primary Completion 2023-08-30 (Actual); Study Completion 2023-08-30 (Actual)

PRIMARY OUTCOMES:
The onset time of sedation | with in 30 minutes before start of surgery
  The onset of sedation will be recorded. It is defined as the time from injection of sedative medications till reaching a target sedation level score 3 by modified Observer's Assessment of Alertness and sedation score (OAA/S).

SECONDARY OUTCOMES:
The extent of airway obstruction | intraopertive
  The extent of airway obstruction by (1= patent airway, 2= airway obstruction alleviated by jaw thrust, 3= airway obstruction alleviated by positive mask ventilation)
rescue analgesic (fentanyl) | intraoperative
  Total number of calling intraoperative rescue analgesic (fentanyl) in both groups will be recorded.
number of participant with complications | intraoperative
  Intraoperative complications such as hypotension (mean arterial blood pressure decreases by > 20% of basal reading), bradycardia (HR decreases by > 20% of basal reading) and bradypnea (RR less than 10 b/m) or hypoxemia (SpO2 less than 95%
Recovery time | with in one hour postoperative
  Recovery time: time from discontinuation of infusion drugs till spontaneous eye opening.
The Neurological status of participants | at baseline then within one hour postoperative
  The Neurological status of participants will be assessed before discharge in the PACU using Markwalder's Neurological Grading scale (MNGs) and recorded:
  Grade 0: no neurologic deficit Grade I: mild symptoms such as headache; absent or mild neurologic deficits such as reflex asymmetry Grade II: drowsiness or disorientation with variable neurologic deficits such as hemiparesis Grade III: stupor, but appropriate responses to noxious stimuli; severe focal signs such as hemiplegia Grade IV: coma with absence of motor response to painful stimuli; decerebrate or decorticate posturing.
surgeon satisfaction | with in 24 hours after surgery
  surgeon satisfaction using 7- point Likert-like verbal rating scale by asking about how they evaluate their experience with anesthetic management during surgery?" score will be 6 and 7 if they are satisfied.5=very satisfied, 4=satisfied, 3= neutral, 2= unsatisfied and 1= very unsatisfied.

CONTACTS AND LOCATIONS:
Overall Officials: Alshaimaa Kamel, M.D, Principal Investigator — Zagazig University
Locations (1):
- Zagazig University Hospitsals, Zagazig, Egypt